CLINICAL TRIAL: NCT04111601
Title: BLI Based Adenoma Surveillance Strategy: BLAST Study
Brief Title: BLI Based Adenoma Surveillance Strategy
Acronym: BLAST
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: King's College Hospital NHS Trust (Other); Luzerner Kantonsspital (Other); Catharina Ziekenhuis Eindhoven (Other); University Medical Centre Ljubljana (Other); Göteborg University (Other); Humanitas Hospital, Italy (Other); Nuovo Regina Margherita Hospital (Other); MITERA Hospitals, Athens , Greece (Unknown)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/30
Record Dates: First submitted 2019-06-12; First posted 2019-10-01 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Blue light imaging — Advanced virtual chromoendoscopy

SUMMARY:
Bowel cancer is the third most common cancer in the UK. It develops through smaller growths in the bowel called polyps. Early recognition and removal of these polyps result in prevention of developing bowel cancer in an individual. However, not all polyps will lead to cancer, certain polyps are just growths of normal tissue and can be left in the bowel. We therefore need to know which polyps to remove and which ones to leave. One way of doing this is to have a better look at these polyps. This can be done by new technologies. One of them is called Blue Light Imaging (BLI). This is a new light source at the end of the camera which is activated by the push of a button. It will help us in looking at these polyps more closely.

This helps us decide which polyps to remove and which ones are safe to leave as there is always a small risk in removing a polyp. It would also give us a better idea as to when to repeat the camera test if necessary (endoscopic surveillance). By reducing the number of polyps resected and sent to the pathology labs for diagnosis, the work load on the pathology department is also reduced and in the process, providing cost savings to the Trust, The study aims to see if using Blue Light during endoscopy helps us to identify and characterize small polyps better

DETAILED DESCRIPTION:
Advanced endoscopic imaging can facilitate the characterisation of neoplastic and non-neoplastic polyps. Accurate identification of small non-neoplastic polyps (e.g. rectosigmoid hyperplastic polyps) that do not harbour malignant potential can lead to future implementation of a 'resect and discard' or 'diagnose and leave' strategy. However, there is insufficient evidence that endoscopists are able to attain high enough levels of optical diagnostic performance in-vivo in order to implement this strategy safely. Blue Light Imaging (BLI) is a new enhanced imaging technology that enhances mucosal surface and vessel patterns. A specific BLI classification was recently developed to enable better characterisation of colorectal polyps (BLI Adenoma Serrated International Classification - BASIC). The use of this technology with the appropriate classification to enhance its performance has not yet been tested in clinical settings of polyp surveillance and screening colonoscopy amongst general endoscopists.

BLAST is a multicentre prospective observational study which will compare BLI optical diagnosis with histological assessment (as a reference standard) for patients with small polyps (<10mm) identified at colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age Able to provide informed consent

Exclusion Criteria:

* History of polyposis syndrome History of Inflammatory bowel disease History of poor bowel prep

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing colonoscopy who fulfill eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage of adenomas correctly identified with BLI | 12 months
  Accuracy of BLI in optical diagnosis of small colorectal polyps

SECONDARY OUTCOMES:
Amount of money saved in GBP ( Cost savings) | 12 months
  Economic implications of replacing histological diagnosis with optical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Z Bhandari, Prof, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospital NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data regarding ensdoscopic findings and histological diagnosis might be shared with other researchers if the need arises.